CLINICAL TRIAL: NCT04654182
Title: Evaluation of the Residual Antimicrobial Efficacy of One Test Material Based on a Modification of ASTM E1115-11 Test Method
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Collaborators: BioScience Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: #2007591-102
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Hand Hygiene
MeSH Terms: interventions — chlorhexidine gluconate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Log reduction in bacterial count (Experimental): Following pre-test period qualifying participants will wash their hands with 4% CHG product 3 times a day over the 5 day study period. Bacterial counts will be taken at 6 and 12 hours after the final wash on day 5 and reductions calculated from the starting count to final count.
  Interventions: Drug: Chlorhexidine Gluconate

INTERVENTIONS:
Drug: Chlorhexidine Gluconate — Product used in accordance with manufacturers Hand Hygiene instructions

SUMMARY:
To evaluate the residual antimicrobial effectiveness of one test product when tested using a modification of the methodology of the standardized ASTM E115-11 (2017)

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be of either sex, between the ages of 18 and 65 years, and of any race.
* Subjects must be able to read and understand English.
* Subjects must possess both hands and all ten digits.
* Subjects must have an average baseline population of at least 1.0 x 105 colony forming units (CFU) per hand.
* Subjects must have no active skin rashes, dermatoses, hangnails, or breaks in the skin of the hands or forearms. Subjects must also have no inflammatory skin conditions, such as dermatitis, eczema, or psoriasis, anywhere on the body.
* Subjects must be in good general health and have no medical diagnosis of a physical condition, such as a current or recent severe illness, a heart murmur, mitral valve prolapse with heart murmur, congenital heart disease, an organ transplant, medicated or uncontrolled diabetes, hepatitis B, hepatitis C, an immunocompromised condition such as AIDS (or HIV positive), lupus, fibromyalgia, ulcerative colitis, Crohn's disease, asthma, heart disease, hypertension, or medicated multiple sclerosis.
* Subjects must have read and signed the Informed Consent Form, List of Restricted Products, and Allowed and Restricted Products For Hand Cleaning During Coronavirus Disease 2019 (COVID-19) Pandemic prior to participating in the study, all located in the separate Informed Consent documents. Subjects must also have a current Authorization to Use and Disclose Protected Health Information Form on file at the testing facility.

Exclusion Criteria:

* Have participated in a clinical study in the past 7 days or be currently participating in another clinical study.
* Wash the hands or applying lotion within the 2-hour period prior to baseline sampling or testing.
* Be experiencing any signs/symptoms of respiratory illness, including cough, fever (body temperature of ≥ 100.0 °F) or chills, shortness of breath or difficulty breathing, persistent pain or pressure in the chest, confusion or inability to respond to external stimuli, bluish lips/face, loss of taste/smell, sore throat, headache, nasal discharge ("runny nose"), frequent sneezing, or general fatigue / body aches.
* Have a current diagnosis of active Coronavirus Disease 2019 (COVID-19) or have been in close contact within the last 2 weeks of anyone who has been diagnosed as having contracted COVID-19.
* Have been regularly smoking or vaping over the past 2 years.
* Have limited mobility or dexterity that would hamper their ability to perform the study as directed.
* Have known allergies or sensitivities to latex (rubber), alcohols, sunscreens, deodorants, laundry detergents, topically applied fragrances, cleansers, soaps, lotions, or to common antibacterial agents, particularly chlorohexidine gluconate.
* Have experienced hives (raised welts) as a reaction to anything that contacted the skin with the exception of plants known to cause reactions for most humans (e.g., poison oak or poison ivy).
* Have a history of anaphylactic shock, anaphylactoid reaction, or anaphylactoid shock.
* Have a known hypersensitivity to the test product or any of its components, especially in those with a history of possible chlorhexidine-related allergic reactions.
* Contact the brain, cerebral membrane, middle ear and eyes with the test product and such contact must be avoided.
* Be receiving any antibiotic medications during the 7-day pre-test period through completion of the study.
* Be receiving any steroids (including steroid medications used to treat asthma) other than for contraception, hormone therapy, or menopausal purposes during the 7-day pre-test period through completion of the study.
* Have any type of port (or portacath) or Peripherally Inserted Central Catheter (PICC).
* Be nursing a child.
* Be pregnant, plan to become pregnant or impregnate a sexual partner within the pre-test and test periods of the study.
* Have any medical condition or use any medications that, in the opinion of the Principal Investigator, or Consulting Physician(s) should preclude participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Bacterial counts | at 6 hours
  Average Log reduction in counts
Bacterial Counts | at 12 hours
  Average Log reduction in counts

CONTACTS AND LOCATIONS:
Locations (1):
- Bioscience Laboratories, Inc, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No